CLINICAL TRIAL: NCT06428877
Title: Monocentric Retrospective Observational Study; Analysis of Gore Excluder ACS Device Using Numerical Simulation
Acronym: ACSSim
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0514
Record Dates: First submitted 2024-05-16; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Vascular Diseases; Surgery
Keywords: Endoprosthesis; Numerical simulation; Proximal neck
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent EVAR with ACS Gore excluder.: Patients who underwent EVAR with ACS Gore excluder. Only patients with proximal neck angulation superior to 60 degrees will be considered.
  Interventions: Other: analyzed on the post-operative scanner

INTERVENTIONS:
Other: analyzed on the post-operative scanner — analyzed on the post-operative scanner

SUMMARY:
andated when the risk of rupture is low and interventional treatment is offered to patients at high risk of rupture. Rupture risk is driven by aneurysm diameter and growth rate. Aneurysms with diameter greater than 55 mm and/or growth rate greater than 1 cm per year are at high risk of rupture. Open surgery and endovascular treatment are the two types of interventions. Open repair consists in replacing the aneurysmal part of the aorta using a synthetic fabric prosthesis after the abdomen has been opened and the aorta clamped. This invasive procedure is associated with a 3-10% post-operative mortality. Endovascular repair (EVAR) consists in excluding the aneurysm sac by inserting a self-expanding prosthesis (called stent-graft) through very small groin incisions, without abdominal opening nor aortic clamping. This minimally invasive procedure is associated with a significantly reduced post-operative mortality (around 1%) . However, hostile proximal neck anatomy including high angulation is associated with higher rates of type IA endoleak, reintervention and long-term mortality . For this reason, a conformable design of the Excluder stent-graft has been engineered with initial satisfactory results in patients with highly angulated or short necks . However, these satisfactory results have been obtained in carefully selected patients from experienced centers and a tool demonstrating adequate apposition of the Gore ACS is lacking. Study Device Description Numerical simulation has been used successfully to predict stent-graft behavior during FEVAR . Preliminary studies have also demonstrated to applicability of the technology to standard infrarenal devices , including in the setting of very tortuous anatomies9 . The potential of numerical simulation to predict stent-graft apposition of Gore ACS in highly angulated necks appears very promising to enhance patient selection.

ELIGIBILITY:
Inclusion Criteria:

The patient:

1. Is age ≥18 at the time of inclusion.
2. Underwent EVAR with ACS Gore Excluder
3. AAA proximal neck angulation superior to 60 degrees
4. Pre-op CT and post-operative/follow-up CT available

Exclusion Criteria:

1. Slice thickness of Pre-op or post-op / follow-up CT superior to 2mm.
2. Non-injected or poorly injected pre-operative CT-scan precluding technical feasibility of the aortic digital twin
3. Absence of post-operative or follow-up CT-scan
4. Patient refusal of his personal information/medical data to be used in the context of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent EVAR with ACS Gore excluder. Only patients with proximal neck angulation superior to 60 degrees will be considered.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The aim of the present study is to investigate the accuracy of numerical simulation to predict stent-graft apposition of Gore ACS in highly angulated proximal AAA necks. | up to 16 months
  Quantitative neck apposition parameters (including but not limited to malapposition length, width, angle) will be extracted both from numerical simulation and post-operative CT.
  Quantitative values will then be compared Comparison between quantitative neck apposition parameters (malapposition length, width, angle) derived from simulation and the one observed on post-op CT and/ or follow-up CT

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided